CLINICAL TRIAL: NCT05552404
Title: Trans-nasal Sphenopalatine Ganglion Block Versus Intravenous Aminophylline Injection for Treatment of Postdural Puncture Headache After Caesarean Section Under Spinal Anesthesia
Brief Title: Postdural Puncture Headache Relief With Aminophylline and SPGB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tamer Samir Abdelsalam, lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU R 124/ 2022
Record Dates: First submitted 2022-09-16; First posted 2022-09-23 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Anesthesia
MeSH Terms: interventions — Conservative Treatment; Aminophylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conservative therapy (Other): will receive conservative therapy such as bed rest, fluids, abdominal binder, oral paracetamol, and caffeine
  Interventions: Other: conservative therapy
- Aminophylline (Active Comparator): will receive conservative therapy plus Aminophylline (250mg of Aminophylline dissolved in 100ml normal saline for intravenous infusion over 30 minutes)
  Interventions: Other: conservative therapy; Drug: Aminophylline
- transnasal spheno-palatine ganglion block (Active Comparator): will receive the conservative therapy plus transnasal spheno-palatine ganglion block under strict protective and safety measures against COVID-19, using a hollow cotton swab soaked in lidocaine 2% for 5 minutes in each nostril then 0.5ml of lidocaine 2% will be injected slowly through the hollow swab and repeated once after another 5 minutes where the patient will stay in the supine position for 10 minutes.
  Interventions: Other: conservative therapy; Procedure: trans nasal sphenopalatine ganglion block

INTERVENTIONS:
Other: conservative therapy — bed rest, fluids, abdominal binder, oral paracetamol, and caffeine
Drug: Aminophylline — conservative therapy plus Aminophylline (250mg of Aminophylline dissolved in 100ml normal saline for intravenous infusion over 30 minutes)
  Arms: Aminophylline
Procedure: trans nasal sphenopalatine ganglion block — conservative therapy plus sphenopalatine ganglion block SPGB using hollow cotton swab and lidocaine 2%
  Arms: transnasal spheno-palatine ganglion block

SUMMARY:
The purpose of the study is to compare Sphenopalatine ganglion block (SPGB) and aminophylline in the efficacy and safety management of PDPH.

DETAILED DESCRIPTION:
Postdural puncture headache (PDPH) is a severe and debilitating complication after regional anesthesia in the obstetric population; The gold standard treatment for PDPH is epidural blood patch, which is an invasive and risky procedure.

The trans-nasal sphenopalatine ganglion (SPG) block and intravenous aminophylline are promising options for PDPH. So the investigators designed this randomized, double-blind study to compare Sphenopalatine ganglion block (SPGB) and aminophylline in the efficacy and safety management of PDPH.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 40 years old female.
* ASA I -II according to the American society of anesthesiologists.
* Spinal anesthesia with 22G Quincke needle for cesarean section.
* PDPH was defined according to the international classification of headache disorders, 3rd edition criteria (ICHD-3) as:

  * Headache occurring within 5 days of a lumbar puncture.
  * Orthostatic headache that significantly worsens soon after sitting upright or standing and/or improves after lying horizontally usually accompanied by neck pain, tinnitus, changes in hearing, photophobia, and/or nausea.
  * Exclusion of other causes such as hypertension, preeclampsia, tension headache, migraine, etc.

Exclusion Criteria:

* A history of headaches that could interfere with the PDPH diagnosis,
* A history of central nervous system diseases, including intracranial hemorrhage, seizures, intracranial hypertension, or hydrocephalus
* A history of cardiovascular diseases, including coronary heart disease, arrhythmias, or hypertension.
* A history of allergy to or any contraindication for using Aminophylline.
* Coagulopathy.
* Nasal septal deviation, polyp, or nasal bleeding.
* General anesthesia after failed spinal anesthesia.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Obstetric participant
Enrollment: 75 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
the headache severity in the form of Visual Analogue score (VAS) at 12 hours after treatment. | at 12 hours
  0 - no pain to 10 - worst pain imaginable

SECONDARY OUTCOMES:
Patient Global impression of change (PGIC) scale | at 24 hours
  Participant encircles number that match degree of change since the begining of care where 0- much better to 10- much worse and 5- no change.
Adverse effects | at 24 hours
  Recording of adverse effects arrhythmias, agitation, and nasal bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: tamer S abdelaziz, MD, Principal Investigator — Faculty of medicine, Ain Shams University, Cairo, Egypt
Locations (1):
- faculty of medicine, Ain Shams University, Cairo, Egypt